CLINICAL TRIAL: NCT05951426
Title: A Study Without a Protocol Number. Documentation Filed in the Registry Under Number 01/19/1438. Date: 08.04.2019.
Brief Title: Expression Analysis of the COPB 2 and Bcl-2 in Early Stages of Endometrial Carcinoma
Status: Completed | Type: Observational
Sponsor: Clinical Center Kragujevac (Other)
Responsible Party: Principal Investigator, Branko Andric, Principal investigator, Clinical Center Kragujevac
Other Study IDs: 01119-1592
Record Dates: First submitted 2023-06-22; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Endometrial Carcinoma Cellular Diagnosis
Keywords: Carcinoma endometrii; apoptosis; relative expression COPB2; relative expression BCL-2; Polymerase Chain Reaction
MeSH Terms: interventions — Ovariectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: 40 patients in whom Endometrial carcinoma was diagnosed as part of the experimental group.
  Interventions: Procedure: 1.hysterectomy with bilateral oophorectomy and pelvic lymphonodectomy. 2 explorative curettage
- control group: 20 patients in whom cancer or atypical hyperplasia of the endometrium was excluded histopathologically.
  Interventions: Procedure: 1.hysterectomy with bilateral oophorectomy and pelvic lymphonodectomy. 2 explorative curettage

INTERVENTIONS:
Procedure: 1.hysterectomy with bilateral oophorectomy and pelvic lymphonodectomy. 2 explorative curettage — 1. removal of the uterus with both ovaries and fallopian tubes and pelvic lymph nodes
  2. exploration of the uterine cavity and removal of the endometrium

SUMMARY:
COPB2 is a subunit of the intracellular transport system between cell organelles that participates in the regulation of cell division and differentiation. Bcl-2 is a protein that participates in regulating the process of apoptosis. Through the research,investigators tried to examine and establish the correlation of the expression of these two genes in endometrial cancer at an early stage.

DETAILED DESCRIPTION:
The research was conducted as a prospective controlled clinical experimental study in the period from 2019-2022. in patients who were treated at the Gynecology and Obstetrics Clinic in Clinical Center Kragujevac. Sections of tissue deriving from the exploratory curettage and operative procedure were taken after obtaining informed consent of participants with the declaration of Helsinki and recommendations of the World Health Organization for experiments on human material and after getting approval of the Ethics Committee.

Participants are divided into two groups. Investigators stored the sample (endometrial tissue) in liquid nitrogen under adequate conditions at the Kragujevac Clinical Center, department for Gynecology and Obstetrics and examined the expression of the COPB2 and Bcl-2 gene in endometrial tissue cells of these two groups of patients. In order to examine the relative expression of the gene for the COPB2 subunit and Bcl-2, investigators sampled endometrial tissue from patients with endometrial cancer - experimental group and from patients without cancer - control group. All participants of the experimental group had initial stages of cancer, without the existence of metastases at the time of taking the sample for the study. Gene expression was performed using the Polymerase Chain Reaction method at the Faculty of Science and Mathematics in Kragujevac.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent of the patient
* pathohistological confirmation of endometrial carcinoma for the experimental group
* normal endometrial tissue and hyperplasia simplex endometrii for the control group.

Exclusion Criteria:

* malignant disease in the patient whose treatment is still ongoing
* pathohistological determination of atypical hyperplasia of the endometrial tissue

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The research was conducted in female patients who were treated at the Gynecology and Obstetrics Clinic in Clinical Center Kragujevac after obtaining informed consent of patients with the declaration of Helsinki and recommendations of the World Health Organization for experiments on human material and after getting approval of the Ethics Committee.
  Female patients are divided into two groups:
  I (first): 40 patients in whom endometrial carcinoma was diagnosed as part of the experimental group and II (second) 20 patients in whom cancer or atypical hyperplasia of the endometrium was excluded histopathologically.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Relative expression COPB2 and BCL-2 | The laboratory processing of the material lasted 3 months, after all the samples were collected during the clinical part of the research. In the period from 01.03. 2022-01.06.2022.
  In order to examine the relative expression of the gene for the COPB2 subunit and Bcl-2, investigators sampled endometrial tissue from patients with endometrial cancer - experimental group and from patients without cancer - control group. All patients of the experimental group had initial stages of cancer, without the existence of metastases at the time of taking the sample for the study. Gene expression was performed using the Polymerase Chain Reaction method

CONTACTS AND LOCATIONS:
Overall Officials: Branko Andrić, MD, Principal Investigator — Department for women's health care, Health Center Raska, Serbia